CLINICAL TRIAL: NCT05937581
Title: A Phase 1, Double-Blind (Sponsor-Unblinded), Placebo-Controlled, Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Single And Multiple Doses Of CSL040 In Healthy Adult Subjects
Brief Title: First-In-Human Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Escalating Single And Multiple Doses Of CSL040 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL040_1001
Record Dates: First submitted 2023-05-18; First posted 2023-07-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Complement-mediated Disorders
Keywords: Complement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part A [Single ascending dose (SAD)]: CSL040 (minimum dose) (Experimental): Single Intravenous (IV) Administration
  Interventions: Drug: CSL040
- Part A (SAD): CSL040 (lower dose) (Experimental): Single IV Administration
  Interventions: Drug: CSL040
- Part A (SAD): CSL040 (low dose) (Experimental): Single IV Administration
  Interventions: Drug: CSL040
- Part A (SAD): CSL040 (medium dose) (Experimental): Single IV Administration
  Interventions: Drug: CSL040
- Part A (SAD): CSL040 (medium-high dose) (Experimental): Single IV Administration
  Interventions: Drug: CSL040
- Part A (SAD): CSL040 (maximum dose) (Experimental): Single IV Administration
  Interventions: Drug: CSL040
- Part A (SAD): Placebo (Placebo Comparator): Single IV Administration
  Interventions: Drug: Placebo
- Part B [Multiple ascending dose (MAD)]: CSL040 (minimum dose) (Experimental): IV Administration not to exceed 5 doses over 14 days
  Interventions: Drug: CSL040
- Part B (MAD): CSL040 (medium dose) (Experimental): IV Administration not to exceed 5 doses over 14 days
  Interventions: Drug: CSL040
- Part B (MAD): CSL040 (high dose) (Experimental): IV Administration not to exceed 5 doses over 14 days
  Interventions: Drug: CSL040
- Part B (MAD): Placebo (Placebo Comparator): IV Administration not to exceed 5 doses over 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CSL040 — IV Administration
  Arms: Part A (SAD): CSL040 (low dose); Part A (SAD): CSL040 (lower dose); Part A (SAD): CSL040 (maximum dose); Part A (SAD): CSL040 (medium dose); Part A (SAD): CSL040 (medium-high dose); Part A [Single ascending dose (SAD)]: CSL040 (minimum dose); Part B (MAD): CSL040 (high dose); Part B (MAD): CSL040 (medium dose); Part B [Multiple ascending dose (MAD)]: CSL040 (minimum dose)
Drug: Placebo — 0.9% w/v NaCI, IV Administration
  Arms: Part A (SAD): Placebo; Part B (MAD): Placebo

SUMMARY:
First-In-Human Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Escalating Single And Multiple Doses Of CSL040 In Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female 18 to 64 years of age, inclusive, at Screening
* 2.Body weight in the range of greater than or equal to (≥) 50 kg and less than or equal to (≤) 100 kilogram (kg) , with a body mass index of ≥ 18 kilogram per meter square (kg/m2) and ≤ 30 kg/m2, at Screening
* 3.Judged as healthy by an Investigator after completion of a comprehensive clinical assessment
* 4.Capable of providing written informed consent and willing and able to adhere to all protocol requirements
* 5.Can understand the nature, scope, and possible consequences of the study and able to comply with study procedures, restrictions, and requirements
* 6. Able to provide proof of adequate vaccination (as determined by the Investigator) against meningococcal disease, including vaccination against meningococcal serogroup B and meningococcal serogroups A, C, W, and Y OR be willing to receive additional vaccinations against these serogroups per the Australian Immunisation Handbook
* 7.Continuous nonsmoker who has not used nicotine- and tobacco-containing products for at least 30 days prior to the first dosing based on urine cotinine testing at Screening and Day-1
* 8.Able to provide proof of adequate vaccination (as determined by the Investigator) against Haemophilus influenzae type b, Pneumococcus OR be willing to receive additional vaccinations against these pathogens with the first dose at least 21 days before the first dose of CSL040
* 9.Able to provide proof of adequate vaccination (as determined by the Investigator) against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS_CoV-2) OR be willing to receive additional vaccination(s) to achieve adequate vaccination status at least 14 days before the first dose of CSL040. If there is proof of a recent SARS-CoV-2 infection (as determined by the Investigator) within 90 days of the first dose of CSL040, the requirement for a vaccination will follow the current local clinical practice

Exclusion Criteria:

* 1.Any individual at high risk of exposure to Neisseria meningitidis, including, but not limited to, health care workers, doctors, nurses, students working in a clinical setting, laboratory workers with exposure to N. meningitidis, individuals residing in a dormitory setting (eg, military workers), and childcare workers
* 2. Vaccination with any live replication-competent vaccine 90 days before Day 1 or planned vaccination with the same within 90 days after the last administration of CSL040
* 3.A positive test result for any of the following: hepatitis B screening, hepatitis C virus antibody, or human immunodeficiency virus-1/2 antibody
* 4.History concerning for a N. meningitidis infection
* 5.History of allergy or intolerance to Penicillin V, as well as to potential backup medications including azithromycin, ciprofloxacin, and ceftriaxone
* 6.History of unexplained, recurrent infection, life-threatening infection, or history that suggests any immunodeficiency (functional immunodeficiency), including asplenia / functional asplenia
* 7.Infection requiring treatment with systemic antibiotics (IV and / or oral administration for more than 3 days) within the last 90 days prior to dosing
* 8.Clinical evidence of current active serious infection, including any localized infection, or any infection which makes participation in this study unacceptably high risk
* 9.Blood pressure or pulse rate measurements outside the normal range for the subject's age and assessed as clinically significant
* 10.Known history of severe hypersensitivity reactions or suspected hypersensitivity to CSL040 or any excipients including polysorbate 80, monoclonal antibodies, or any documented history of a severe allergic reaction (in the opinion of the Investigator), angioedema, or anaphylaxis to food or any other drugs.
* 11.Subject has any condition that may compromise their safety or compliance, impede successful conduct of the study, interfere with interpretation of the results or would otherwise render the subject unsuitable for participation in the study
* 12.A positive test result for drugs of abuse (including alcohol) and cotinine at Screening and / or Day -1.
* 13.Weekly alcohol intake of > 10 units for females and > 14 units for males during the 3 months before Day -1.
* 14.Any values above the upper limit of normal (ULN) for alanine aminotransaminase (ALT) or aspartate aminotransaminase (AST), or bilirubin test result
* 15.Use of prescription or over-the-counter medication, herbal and dietary supplements, and vitamins and minerals (except any vaccinations or other medications required/permitted as per protocol) within the 21 days before first administration of investigational product
* 16.Female subject of childbearing potential or fertile male subject who are neither using nor willing to use a highly effective method of contraception
* 17.Pregnant, lactating, or breastfeeding
* 18.Donation or loss of more than 500 milliLiter (mL) of blood within 3 months, or donation of plasma within 7 days, before admission to the unit or plans to donate blood or plasma and for 5 half-lives of the last dose of CSL040 or until the end of the study, whichever is longer
* 19.Any planned surgical procedures during the study period
* 20.Participation in any other investigational product study in which receipt of an investigational product occurred within 5 half-lives or 28 days (whichever is longer) before dosing of investigational product, or participation in more than 4 clinical studies involving administration of an investigational product within the last 12 months before Screening
* 21.Subject who met all eligibility criteria but was not needed (ie, alternate subjects). Alternate subjects are eligible to participate in subsequent cohorts
* 22. Prior dosing with CSL040

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs), adverse events of special interests (AESIs), and serious adverse events (SAEs) | Part A (SAD): Up to 105 days; Part B (MAD): Up to 174 days
Percentages of participants with TEAEs, AESIs, and SAEs | Part A (SAD): Up to 105 days; Part B (MAD): Up to 174 days
The Number of Clinically Significant Changes from Baseline in Clinical Laboratory Tests Reported as AE | Baseline and up to 69 days
  Clinical laboratory tests include hematology, biochemistry, coagulation, and urinalysis collected during the study. The investigator determines if the changes in laboratory test results are clinically significant.
Number of participants with vital signs out of normal range | Baseline and up to 69 days
  Blood pressure (systolic and diastolic), pulse rate, respiratory rate and tympanic temperature will be assessed.
Change from Baseline in corrected QT interval using Fridericia's formula (QTcF) values of triplicate electrocardiograms | Baseline and up to 69 days
Absolute values of QTcF on electrocardiograms | Baseline and up to 69 days
Number of participants with abnormal electrocardiogram findings | Baseline and up to 69 days

SECONDARY OUTCOMES:
Part A (SAD): Maximum concentration (Cmax) | Up to 56 days
Part A (SAD): Time to reach maximum concentration (Tmax) | Up to 56 days
Part A (SAD): Time to Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-last) | Up to 56 days
Part A (SAD): Area under the concentration-time curve from time 0 to infinity (AUC0-infinity) | Up to 56 days
Part A (SAD): Total systemic clearance (CL) | Up to 56 days
Part A (SAD): Volume of distribution (V) | Up to 56 days
Part A (SAD): Terminal elimination half-life (T1/2) | Up to 56 days
Part B (MAD): Maximum concentration (Cmax) | Up to 69 days
Part B (MAD): Time to reach maximum concentration (Tmax) | Up to 69 days
Part B (MAD): Time to Area under the concentration-time curve in 1 dosing interval (AUCtau) | Up to 69 days
Part B (MAD): Accumulation index (accumulation ratio determined by the ratio of steady state AUCtau to single dose AUCtau) | Up to 69 days
Part B (MAD): Lowest concentration prior to dosing (Ctrough) | Up to 69 days
Part B (MAD): Total systemic clearance (CL) | Up to 69 days
Part B (MAD): Volume of distribution at steady state (Vss) | Up to 69 days
Part A (SAD) and Part B (MAD): Percent change from Baseline in pharmacodynamic (PD) parameters | Up to 56 days (Part A) and up to 69 days (Part B)
  Levels of Wieslab ex vivo pathway activity for classical, lectin and alternative complement pathways, CH50 (hemolysis of sheep erythrocytes) and ApH50 (hemolysis of rabbit erythrocytes) will be measured and for each PD parameter presented as percent change from baseline over time profiles.
Part A (SAD) and Part B (MAD): Maximum percent change from Baseline (Emax) in PD parameters | Up to 56 days (Part A) and up to 69 days (Part B)
  Levels of Wieslab ex vivo pathway activity for classical, lectin and alternative complement pathways, CH50 and ApH50 will be measured and for each PD parameter the maximum percent change from Baseline (Emax) will be determined.
Part A (SAD) and Part B (MAD): Time to maximum percent change from Baseline (TEmax) in PD parameters | Up to 56 days (Part A) and up to 69 days (Part B)
  Levels of Wieslab ex vivo pathway activity for classical, lectin and alternative complement pathways, CH50 and ApH50 will be measured and for each PD parameter the Time to maximum percent change from Baseline (TEmax) will be determined.
Part A (SAD) and Part B (MAD): Time below Baseline in PD parameters | Up to 56 days (Part A) and up to 69 days (Part B)
  Levels of Wieslab ex vivo pathway activity for classical, lectin and alternative complement pathways, CH50 and ApH50 will be measured and for each PD parameter the Time below Baseline will be determined.
Part A (SAD) and Part B (MAD): AUC below Baseline in PD parameters | Up to 56 days (Part A) and up to 69 days (Part B)
  Levels of Wieslab ex vivo pathway activity for classical, lectin and alternative complement pathways, CH50 and ApH50 will be measured and for each PD parameter the AUC below Baseline will be determined.
Part A (SAD) and Part B (MAD): Number of serum samples with Positive antidrug antibodies (ADAs) binding to CSL040 | Up to 56 days (Part A) and up to 69 days (Part B)
Part A (SAD) and Part B (MAD): Number of participants with presence of treatment-emergent ADAs | Up to 56 days (Part A) and up to 69 days (Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSLBehring LLC
Locations (1):
- Nucleus Network Pty Ltd, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e. FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.